CLINICAL TRIAL: NCT05850806
Title: Effectiveness, Acceptability and Feasibility of "KmAsthma" Self-management App in iMprovIng the ContRol Of aSthma (MICROS) Among Day Scholar Secondary School Adolescents in Kampala City Uganda: A Cluster Randomised Controlled Trial
Brief Title: Effectiveness of a Self-management App in Improving the Control of Asthma Among School Adolescents
Acronym: MICROS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Mak-SOMREC-2021-67
Record Dates: First submitted 2023-04-29; First posted 2023-05-09 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Asthma
Keywords: Asthma control; KmAsthma; Phone app; Adolescents; School; Low resource settings
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants and the assessors will be masked to the study arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KmAsthma self-management smart phone app intervention (Experimental): Participants assigned to the intervention arm will be given a link to download the self-management app on their Android smartphone or iPhone
  Interventions: Device: The KmAsthma self-management smart phone app intervention
- Control arm (No Intervention): Will emulate standard access to asthma self-management information

INTERVENTIONS:
Device: The KmAsthma self-management smart phone app intervention — KmAsthma is a free app which enables users to track their symptoms, access their action plan, learn about asthma and set goals to make change
  Arms: KmAsthma self-management smart phone app intervention

SUMMARY:
Uganda experiences high morbidity and costs due to uncontrolled asthma. Poor asthma control in adolescents is partly attributed to inadequate asthma education; indicating that education and self-management programs are essential components of asthma control. Adolescents with poorly controlled asthma are reported to have improved asthma control after using a smart phone application in outpatient setting studies. However, there is paucity of data on the effectiveness, feasibility and acceptability of smart phone applications in the control of asthma among adolescent secondary school students in low resource settings.

DETAILED DESCRIPTION:
Uganda experiences high morbidity and costs due to uncontrolled asthma. Poor asthma control in adolescents is partly attributed to inadequate asthma education; indicating that education and self-management programs are essential components of asthma control. Adolescents with poorly controlled asthma are reported to have improved asthma control after using a smart phone application in outpatient setting studies. However, there is paucity of data on the effectiveness, feasibility and acceptability of smart phone applications in the control of asthma among adolescent secondary school students in low resource settings. This study will evaluate the effectiveness, acceptability and feasibility of the "KmAsthma" self-management app in improving the control of asthma among day scholar secondary school adolescents in Kampala City Uganda.

This study is a 6-month cluster randomized, controlled, single-centre, single-blinded, pragmatic parallel trial, with two arms and a primary endpoint of improving the control of uncontrolled asthma measured as change in individual mean scores on the Asthma control questionnaire during a self-management intervention delivered by the "KmAsthma" smartphone app. The study will compare students with uncontrolled asthma in the intervention group using the "KmAsthma" smartphone app (T) with the students in the control arm (C) who will receive no intervention. Data will be analysed by summarizing descriptive statistics; determining odds ratios for asthma control using logistic regression models, using repeated measures ANCOVA for repeated continuous measurements. Permission from CEU and approval from SOMREC and UNCST will be sought. Informed and written consent and assent will sought. Dissemination will be through publications and presentations in local and international conferences. The findings may contribute to filling the gap leading to overall unsatisfactory asthma control in adolescents.

ELIGIBILITY:
Inclusion Criteria for Schools:

* Secondary schools in Kampala
* School has existed for more than five years

Exclusion criteria for schools:

* Schools already participating in an asthma related randomised controlled trial

Inclusion criteria for students:

* 12-19 years
* Day scholar student
* Uncontrolled asthma on assessment using Asthma Control Test (ACT score less than 19)
* Self-reported access to a smart phone

Exclusion criteria for students:

* Students already taking part in an asthma-related randomised controlled trial
* Too sick to use the smart phone

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Change in mean Asthma Control Test (ACT) scores | Baseline, 3 and 6 months
  The ACT questionnaire is composed of five questions, each scored on a scale from 1 to 5, with a total score range of 5 to 25. A score of 19 or above is considered indicative of well-controlled asthma

SECONDARY OUTCOMES:
Adolescent Asthma Self-Efficacy Questionnaire (AASEQ) | Baseline, 3 and 6 months
  Change in AASEQ scores
Feasibility based on proportion of participants that will drop out of the study | Baseline, 3 and 6 months
  Deemed feasible if the percentage of participants who drop out of the study (i.e., fail to complete any of the tools) is less than 15%

CONTACTS AND LOCATIONS:
Overall Officials: James Davis Katumba, MSc, Principal Investigator — Makerere University, College of Health Sciences, Clinical Epidemiology Unit

IPD SHARING:
Plan to Share IPD: Yes
All the individual participant data collected after de-identification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication
Access Criteria: Data available indefinitely at the link that will be added
URL: https://orcid.org/0000-0001-8617-3786

REFERENCES:
- [Background] Nathan RA, Sorkness CA, Kosinski M, Schatz M, Li JT, Marcus P, Murray JJ, Pendergraft TB. Development of the asthma control test: a survey for assessing asthma control. J Allergy Clin Immunol. 2004 Jan;113(1):59-65. doi: 10.1016/j.jaci.2003.09.008. PMID 14713908
- [Background] Holley S, Knibb R, Latter S, Liossi C, Mitchell F, Radley R, Roberts G. Development and validation of the Adolescent Asthma Self-Efficacy Questionnaire (AASEQ). Eur Respir J. 2019 Jul 4;54(1):1801375. doi: 10.1183/13993003.01375-2018. Print 2019 Jul. PMID 31048348
- [Result] Davis SR, Peters D, Calvo RA, Sawyer SM, Foster JM, Smith L. "Kiss myAsthma": Using a participatory design approach to develop a self-management app with young people with asthma. J Asthma. 2018 Sep;55(9):1018-1027. doi: 10.1080/02770903.2017.1388391. Epub 2017 Nov 28. PMID 29064746
- [Derived] Katumba JD, Kirenga B, Muwagga Mugagga A, Kalyango JN, Nantanda R, Karamagi C. MICROS: Asthma Control App for School Adolescents in a Low Resource Setting - A Cluster Randomized Controlled Trial Protocol. Patient Prefer Adherence. 2023 Nov 30;17:3125-3133. doi: 10.2147/PPA.S438549. eCollection 2023. PMID 38053534